CLINICAL TRIAL: NCT02363868
Title: Costs and Outcome Among Patients With Chronic Myelogenous Leukemia (CML) Receiving Dasatinib or Nilotinib as First or Second Line Therapy in a Commercial and Medicare Population
Brief Title: Healthcare Costs Among Patients With CML Receiving Dasatinib or Nilotinib in a Commercial and Medicare Population
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-568
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CML subjects receiving Dasatinib: CML receiving dasatinib as first or second line therapy will be conducted to assess healthcare costs
- CML subjects receiving Nilotinib: CML receiving nilotinib as first or second line therapy will be conducted to assess healthcare costs

SUMMARY:
The purpose of this study is to examine the healthcare costs among patients with CML receiving dasatinib or nilotinib as first line therapy in a commercially or Medicare insured population.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Age >18 years
* International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9 CM) code for CML (205.1x)
* At least 2 prescriptions for dasatinib or nilotinib from July 1, 2008 to June 31, 2013
* Continuous eligibility for the 6 months pre- and post-index date (defined as the date of first fill for dasatinib or nilotinib)

Exclusion Criteria:

* History of bone marrow or stem cell transplant as identified in the 6 month pre-period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Others: Retrospecitve database analysis of patients in a health plan
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Healthcare costs | Intent-to-treat (ITT) at 6 months
  Average (mean) costs for patients receiving dasatinib or nilotinib as first line therapy

SECONDARY OUTCOMES:
Healthcare costs by line of therapy | Intent-to-treat (ITT) at 6 months
Resource utilization by line of therapy | Intent-to-treat (ITT) at 6 months
  Captured per number of hospitalizations, Emergency room (ER) visits, physician office visits, and medications / number of prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Franklin Pharmaceutical Consulting, Llc, Clinton, South Carolina, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx